CLINICAL TRIAL: NCT00112489
Title: A Phase II Evaluation of Paclitaxel (Taxol, NSC # 673089) and Carboplatin (Paraplatin, NSC #241240) in the Treatment of Advanced, Persistent, or Recurrent Uterine Carcinosarcoma
Brief Title: Paclitaxel and Carboplatin in Treating Patients With Persistent or Recurrent Stage III or Stage IV Uterine Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000432956; GOG-0232B
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2014-04

CONDITIONS: Sarcoma
Keywords: recurrent uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; uterine carcinosarcoma
MeSH Terms: conditions — Sarcoma | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Taxol-Carbo (Experimental): Paclitaxel 175 mg/m2 IV over 3 hours followed by carboplatin AUC = 6 IV over 30 minutes every 21 days until disease progression or adverse effects prohibit further therapy
  Interventions: Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving paclitaxel together with carboplatin works in treating patients with persistent or recurrent stage III or stage IV uterine cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of paclitaxel and carboplatin in patients with persistent or recurrent stage III or IV uterine carcinosarcoma.
* Determine the nature and degree of toxicity of this regimen in these patients.

OUTLINE: This is a non-randomized, multicenter study.

Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: Approximately 14-47 patients will be accrued for this study within 20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed uterine carcinosarcoma (mixed mesodermal tumor)

  * Stage III or IV disease
  * Persistent or recurrent disease
* Documented disease progression
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan

  * At least 1 target lesion

    * Tumors within a previously irradiated field are not considered target lesions unless there is documented disease progression
* Ineligible for any higher priority Gynecology Oncology Group (GOG) protocol (i.e., any active GOG phase III protocol for the same patient population)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* GOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No sensory or motor neuropathy > grade 1

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior cytotoxic chemotherapy for uterine sarcoma

Endocrine therapy

* At least 1 week since prior hormonal therapy for uterine sarcoma
* Concurrent hormone replacement therapy allowed

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Other

* Recovered from all prior therapy
* No prior anticancer therapy that would preclude study therapy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2005-05; Primary Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A. Powell, MD, Study Chair — Washington University Siteman Cancer Center
Locations (110):
- United States (99):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - St. Vincent's Medical Center, Jacksonville, Florida
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish St. Peters Hospital - Saint Louis, St Louis, Missouri
  - Saint Mary's Health Center, St Louis, Missouri
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Jersey Shore Cancer Center at Jersey Shore University Medical Center, Neptune City, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Mount Sinai Medical Center, New York, New York
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Piedmont Hematology-Oncology Associates, Winston-Salem, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Midtown Tulsa, Tulsa, Oklahoma
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center CCOP Research Base, Philadelphia, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Black Hills Obstetrics & Gynecology LLP, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Hall and Martin, M.Ds., PC, Knoxville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Carilion Gynecologic Oncology Associates, Roanoke, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Japan (11):
  - Iwate Medical University Hospital, Morioka, Iwate
  - Kagoshima City Hospital, Kagoshima City, Kagoshima
  - Kobe Medical Center, Kobe
  - National Hospital Organization - Medical Center of Kure, Kure
  - Shikoku Cancer Center, Matsuyama
  - National Kyushu Cancer Center, Minamiku
  - Kinki University School of Medicine, Osaka, Osaka
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Graduate School of Medicine, Sendai
  - Keio University School of Medicine, Shinjuku-ku
  - Tottori University Hospital, Tottori

REFERENCES:
- [Result] Powell MA, Filiaci VL, Rose PG, Mannel RS, Hanjani P, Degeest K, Miller BE, Susumu N, Ueland FR. Phase II evaluation of paclitaxel and carboplatin in the treatment of carcinosarcoma of the uterus: a Gynecologic Oncology Group study. J Clin Oncol. 2010 Jun 1;28(16):2727-31. doi: 10.1200/JCO.2009.26.8326. Epub 2010 Apr 26. PMID 20421537

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel Followed by Carboplatin: Paclitaxel 175 mg/m2 IV over 3 hours followed by Carboplatin AUC = 6 IV over 30 minutes repeated every 21 days until disease progression or adverse effects prohibit further therapy
Period: Overall Study
Arm/Group | Paclitaxel Followed by Carboplatin
Started | 55 (All patients enrolled on study)
Completed | 15 (Completed regimen due to progression)
Not Completed | 40
Not completed — Refused further treatment | 8
Not completed — Adverse Event | 12
Not completed — Death | 2
Not completed — Other, Not Specified | 9
Not completed — Patient never treated | 2
Not completed — Ineligible | 7

BASELINE CHARACTERISTICS:
Population: Total eligible and treated participants
Arm/Group | Paclitaxel Followed by Carboplatin
Number analyzed (Participants) | 46
Age, Customized [Mean (Standard Deviation); unit: years]
  Age at Study Entry | 65.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Nature and Degree of Toxicity
Description: Number of patients who experienced grade 1 or higher serious adverse event (term or group) regardless of attribution using CTCAE v3.0
Time Frame: During study treatment and up to 30 days after stopping study treatment
Population: Eligible and Evaluable patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE
- Grade 1 (CTCAE v 3.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 3.0
- Grade 2 (CTCAE v 3.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 3.0
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 3.0
- Grade 4 (CTCAE v 3.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 3.0
- Grade 5 (CTCAE v.3.0): Number of patients who experienced a grade 5 event using Common Terminology Criteria version 3.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v 3.0) | Grade 2 (CTCAE v 3.0) | Grade 3 (CTCAE v 3.0) | Grade 4 (CTCAE v 3.0) | Grade 5 (CTCAE v.3.0)
Number analyzed (Participants) | 46 | 46 | 46 | 46 | 46 | 46
Participants
  Leukopenia | 2 | 4 | 20 | 19 | 1 | 0
  Neutropenia | 1 | 3 | 3 | 19 | 20 | 0
  Thrombocytopenia | 17 | 19 | 5 | 3 | 2 | 0
  Anemia | 4 | 10 | 27 | 3 | 2 | 0
  Other hematologic | 43 | 0 | 1 | 2 | 0 | 0
  Allergy | 40 | 3 | 0 | 3 | 0 | 0
  Auditory | 43 | 0 | 2 | 1 | 0 | 0
  Cardiovascular | 39 | 3 | 2 | 1 | 1 | 0
  Coagulation | 45 | 0 | 1 | 0 | 0 | 0
  Constitutional | 33 | 8 | 4 | 1 | 0 | 0
  Fatigue | 9 | 14 | 19 | 4 | 0 | 0
  Alopecia | 8 | 7 | 31 | 0 | 0 | 0
  Dermatologic | 36 | 8 | 2 | 0 | 0 | 0
  Endocrine | 44 | 2 | 0 | 0 | 0 | 0
  Gastrointestinal | 18 | 12 | 14 | 2 | 0 | 0
  Nausea | 17 | 20 | 8 | 1 | 0 | 0
  Vomiting | 35 | 7 | 3 | 1 | 0 | 0
  Diarrhea | 35 | 8 | 2 | 1 | 0 | 0
  Stomatitis | 35 | 1 | 0 | 0 | 0 | 0
  Genitourinary/renal | 45 | 1 | 0 | 0 | 0 | 0
  Hemorrhage | 43 | 1 | 2 | 0 | 0 | 0
  Hepatic | 45 | 0 | 0 | 1 | 0 | 0
  Febrile neutropenia | 45 | 0 | 0 | 1 | 0 | 0
  Metabolic | 23 | 18 | 4 | 1 | 0 | 0
  Creatinine | 44 | 2 | 0 | 0 | 0 | 0
  Musculoskeletal | 41 | 2 | 2 | 1 | 0 | 0
  Neurologic | 40 | 0 | 4 | 2 | 0 | 0
  Neuromotor | 44 | 0 | 2 | 0 | 0 | 0
  Sensory neuropathy | 14 | 15 | 12 | 5 | 0 | 0
  Ocular/visual | 43 | 2 | 1 | 0 | 0 | 0
  Pain | 35 | 3 | 6 | 0 | 2 | 0
  Myalgia | 35 | 3 | 7 | 1 | 0 | 0
  Arthralgia | 36 | 4 | 6 | 0 | 0 | 0
  Pulmonary | 37 | 5 | 2 | 2 | 0 | 0

2. Primary Outcome: Response Evaluation Criteria in Solid Tumors Criteria (RECIST) 1.0 Best Response
Description: Primary outcome measured according to RECIST v1.0 Best Response:
  Complete Response (CR) is disappearance of all target and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart Disease Progression is at least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD or the appearance of new lesions within 8 weeks of study entry.
  Partial Response (PR) is at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of nontarget lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required Stable Disease is any condition not meeting the above criteria. Indeterminate is defined as having no repeat tumor assessments following initiation of study therapy for reasons unrelated to symptoms or signs of disease.
Time Frame: Response was measured every other cycle (q 6 weeks) until disease progression is documented.
Population: Total eligible and treated participants
Measure: Number; unit: participants
Arm/Group | Paclitaxel Followed by Carboplatin
Number analyzed (Participants) | 46
participants
  Complete Response | 6
  Partial Response | 19
  Stable Disease | 11
  Disease Progression | 6
  Indeterminate | 4

ADVERSE EVENTS:
Time Frame: During active treatment and up to 30 days after stopping the study treatment.
Description: Treated & eligible patients. Due to the methods in which Adverse Events(AEs) were collected &/or stored, it is not possible to report only the Other(not including Serious) AEs in the appropriate table. Therefore it is a combined set of SAEs & non-serious AEs. Other AEs are Grade 2 or worse & are restricted to those thought to be treatment related.
Arm/Group | Paclitaxel Followed by Carboplatin
Serious Adverse Events (participants affected / at risk) | 11/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel Followed by Carboplatin (N=46)
PTT (Vascular disorders) | 1
Fatigue (General disorders) | 1
Cardiac ischemia/infarction (Cardiac disorders) | 1
S/n arrhythmia: atrial fibrillation (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 1
Death, no ctcae term - death nos (General disorders) | 1
Death, no ctcae term - disease progression (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Dehydration (Gastrointestinal disorders) | 1
Distention (Gastrointestinal disorders) | 1
Obstruction, gi - colon (Gastrointestinal disorders) | 1
Gastrointestinal - other (Gastrointestinal disorders) | 1
Leukocytes (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Neutrophils (Blood and lymphatic system disorders) | 2
Inf w/nml or gr 1 or 2 anc: urinary tract (Infections and infestations) | 1
Inf unknown anc: bladder (urinary) (Infections and infestations) | 1
Inf unknown anc: urinary tract nos (Infections and infestations) | 1
Muscle weakness - extremity-lower (Musculoskeletal and connective tissue disorders) | 1
muscle weakness - extremity-upper (Musculoskeletal and connective tissue disorders) | 1
Bilirubin (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pain: abdominal pain nos (General disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel Followed by Carboplatin (N=46)
Leukopenia (Blood and lymphatic system disorders) | 40
Neutropenia (Blood and lymphatic system disorders) | 43
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Anemia (Blood and lymphatic system disorders) | 32
Other Hematologic (Blood and lymphatic system disorders) | 3
Allergy (Immune system disorders) | 3
Auditory (Ear and labyrinth disorders) | 3
Cardiovascular (Cardiac disorders) | 4
Coagulation (Vascular disorders) | 1
Constitutional (General disorders) | 5
Fatigue (General disorders) | 24
Alopecia (Skin and subcutaneous tissue disorders) | 31
Dermatologic (Skin and subcutaneous tissue disorders) | 2
Death (General disorders) | 2
Other, Gastrointestinal (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 3
Hemorrhage (Blood and lymphatic system disorders) | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Metabolic (Metabolism and nutrition disorders) | 6
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3
Neurologic (Nervous system disorders) | 6
Neuromotor (Nervous system disorders) | 2
Sensory Neuropathy (Nervous system disorders) | 18
Ocular/Visual (Eye disorders) | 1
Pain (General disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No